CLINICAL TRIAL: NCT01609231
Title: A Phase IIA Open Label, Adaptive, Randomized Clinical Trial of Dalotuzumab (MK-0646) Treatment in Combination With Irinotecan Versus Cetuximab and Irinotecan for Patients With Metastatic Rectal Cancers (mRC) Expressing High IGF-1/Low IGF-2 Levels
Brief Title: A Trial of Dalotuzumab in Combination With Irinotecan Versus Cetuximab and Irinotecan for Participants With Metastatic Rectal Cancers (mRC) (MK-0646-025)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This trial was halted prematurely for business reasons and low enrollment.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0646-025; 2012-000317-36 (EudraCT Number); MK-0646-025 (Other: Merck Protocol Number)
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Results first posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — dalotuzumab; Irinotecan; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Dalotuzumab + Irinotecan (Experimental): Participants receive irinotecan intravenously (IV), 180 mg/m^2 once every two weeks + dalotuzumab IV, 10 mg/kg once weekly, during ≥1 42-day treatment cycle(s).
  Interventions: Drug: Dalotuzumab; Drug: Irinotecan
- Arm B: Cetuximab + Irinotecan (Active Comparator): Participants receive cetuximab IV, initial dose of 400 mg/m^2 and then 250 mg/m^2 IV weekly + irinotecan IV, 180 mg/m^2 once every two weeks, during ≥1 42-day treatment cycle(s).
  Interventions: Drug: Irinotecan; Drug: Cetuximab

INTERVENTIONS:
Drug: Dalotuzumab — Dalotuzumab will be administered intravenously after the completion of irinotecan infusion at a dose of 10 mg/kg once weekly.
  Other Names: MK-0646
  Arms: Arm A: Dalotuzumab + Irinotecan
Drug: Irinotecan — Irinotecan 180 mg/m^2 will be administered intravenously once every two weeks either prior to dalotuzumab (Arm A) or after cetuximab (Arm B). Pre-medication at the discretion of the investigator will follow local or country-specific standard of care.
  Other Names: Camptosar
Drug: Cetuximab — Cetuximab will be administered intravenously prior to irinotecan at an initial dose of 400 mg/m^2 followed by weekly infusions of 250 mg/m^2. Pre-medication at the discretion of the investigator will follow local or country-specific standard of care.
  Other Names: Erbitux
  Arms: Arm B: Cetuximab + Irinotecan

SUMMARY:
The purpose of this adaptive trial is to compare the progression-free survival of participants with metastatic rectal carcinoma when treated with intravenous (IV) dalotuzumab (MK-0646) + irinotecan therapy relative to participants treated with IV cetuximab + irinotecan. The primary hypothesis is that administration of dalotuzumab in combination with irinotecan to participants with wild-type KRAS metastatic rectal carcinoma with high insulin growth factor (IGF)-1/low IGF-2 expression levels improves progression-free survival compared to patients treated with cetuximab in combination with irinotecan.

ELIGIBILITY:
Inclusion Criteria:

* Has metastatic colorectal cancer with primary tumor originating from the rectum
* Has an available archival (recent or remote) tumor, or newly obtained formalin-fixed tissue available for analysis for biomarker studies
* Has at least one measurable lesion greater than or equal to 10 mm
* Disease has progressed after treatment with both irinotecan- and oxaliplatin-containing regimens and should have progressed on or within 3 months of completing their last line of therapy
* Has a performance status 0-1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale

Exclusion Criteria:

* Has poorly-controlled diabetes
* Has received chemotherapy or biological therapy within 2 weeks prior to initial dosing on this study, or whose toxicities from agents administered 2 weeks earlier have not resolved to at least grade 1 or baseline, or who is within 3 weeks from a prior surgery
* Has received radiotherapy within 2 weeks prior to initial dosing on this study, unless the radiotherapy was for management of pain
* Is currently participating or has participated in a study with an investigational compound or device within 30 days or 5 half-lives of the investigational agent, whichever is longer, of initial dosing on this study
* Was unable to complete previous course of irinotecan due to intolerable toxicity, other than discontinuation due to fatigue following prolonged administration (>4 months exposure)
* Has prior exposure to insulin-like growth factor 1 receptor (IGF-1R) inhibitors or epidermal growth factor receptor (EGFR) inhibitors
* Has a known central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has primary CNS tumor
* Has a history of a prior malignancy with the exception of cervical intraepithelial neoplasia; basal cell carcinoma of the skin; adequately treated localized prostate carcinoma; potentially curative therapy with no evidence of that disease for 5 years, deemed low risk for recurrence by treating physician.
* Is human immunodeficiency virus (HIV)-positive
* Has active hepatitis B or C infection and is receiving antiviral treatment regimens
* Has symptomatic ascites or pleural effusion
* Is concurrently using growth hormone (GH), or growth hormone inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-07-06 (Actual); Primary Completion 2014-12-09 (Actual); Study Completion 2014-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was halted prematurely for business reasons.
Groups:
- Dalotuzumab + Irinotecan: Participants received irinotecan intravenously (IV), 180 mg/m^2 once every two weeks + dalotuzumab IV, 10 mg/kg once weekly, during ≥1 42-day treatment cycle(s).
- Cetuximab + Irinotecan: Participants received cetuximab IV, initial dose of 400 mg/m^2 and then 250 mg/m^2 IV weekly + irinotecan IV, 180 mg/m^2 once every two weeks, during ≥1 42-day treatment cycle(s).
Period: Overall Study
Arm/Group | Dalotuzumab + Irinotecan | Cetuximab + Irinotecan
Started | 6 | 5
Completed | 3 | 2
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dalotuzumab + Irinotecan: Participants received irinotecan IV, 180 mg/m^2 once every two weeks + dalotuzumab IV, 10 mg/kg once weekly, during ≥1 42-day treatment cycle(s).
- Total: Total of all reporting groups
Arm/Group | Dalotuzumab + Irinotecan | Cetuximab + Irinotecan | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (13.8) | 64.6 (9.9) | 60.5 (12.3)
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 4 | 1 | 5
  From 65-84 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Progression-free Survival (PFS)
Description: PFS is a measure of the time from randomization to the time of first documented disease progression (assessed by an independent Radiology Review Committee [iRRC]) or participant death, whichever occurs first.
Time Frame: From randomization (Cycle 1, Day 1) to the first documented disease progression or death due to any cause, whichever occurs first (up to 3 years)
Population: Due to low enrollment and early termination of study, insufficient data were collected for this endpoint, and no endpoint data were assessed by the iRRC.
Arm/Group | Dalotuzumab + Irinotecan | Cetuximab + Irinotecan
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Participants With Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants achieving a complete response (CR) or partial response (PR) during the course of the study using enhanced Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Confirmation of response was not required.
Time Frame: as for outcome 1
Population: Due to low enrollment and early termination of study, insufficient data were collected for this endpoint, and no endpoint data were assessed for RECIST 1.1 criteria.
Arm/Group | Dalotuzumab + Irinotecan | Cetuximab + Irinotecan
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 553 days
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participants administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. All randomized participants who received ≥1 dose of study therapy are included in the safety analysis.
Arm/Group | Dalotuzumab + Irinotecan | Cetuximab + Irinotecan
All-Cause Mortality (participants affected / at risk) | 1/6 | 2/5
Serious Adverse Events (participants affected / at risk) | 1/6 | 4/5
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalotuzumab + Irinotecan (N=6) | Cetuximab + Irinotecan (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalotuzumab + Irinotecan (N=6) | Cetuximab + Irinotecan (N=5)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (2)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 6 (23) | 4 (18)
Dry mouth (Gastrointestinal disorders) | 1 (6) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival oedema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (7) | 4 (9)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (6) | 2 (5)
Asthenia (General disorders) | 2 (6) | 1 (4)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (2) | 2 (3)
Mucosal inflammation (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (2) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Gingival abscess (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (3)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (3) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 1 (3)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 4 (16) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Bone erosion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
Circadian rhythm sleep disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (3)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (6)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (6)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study did not meet target enrollment and was terminated for business reasons; insufficient data were collected for efficacy analyses. Safety data are reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.